CLINICAL TRIAL: NCT02905461
Title: A Randomised Controlled Trial of an Intervention Delivered by Text Message to Increase the Acceptability of Effective Contraception Among Young Women in Palestine
Brief Title: An Intervention Delivered by Text Message to Increase the Acceptability of Effective Contraception Among Young Women in Palestine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Palestinian Family Planning and Protection Association (Other); International Planned Parenthood Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10831
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: Reproductive health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Contraceptive text messages
  Interventions: Behavioral: Contraceptive text messages
- Control (Placebo Comparator): Text messages not about contraception
  Interventions: Other: Text messages not about contraception

INTERVENTIONS:
Behavioral: Contraceptive text messages
  Arms: Intervention
Other: Text messages not about contraception
  Arms: Control

SUMMARY:
This randomised controlled trial will establish the effect a contraceptive intervention delivered by mobile phone text message on the acceptability of effective contraception in Palestine. Woman aged 18-24 will be randomised to receive 0-3 text messages a day for 4 months (intervention) or a monthly text message not about contraception (control). Participants will complete a questionnaire at baseline and 4 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24 years
* Own a personal mobile phone
* Not using the pill, implant, injection, intrauterine device or patch
* Live in the West Bank

Exclusion Criteria:

* Cannot read Arabic

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 586 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of at least one method of effective contraception | 4 months
  The proportion reporting that at least one method of effective contraception is acceptable (pill, intrauterine device, injection, implant, patch)

SECONDARY OUTCOMES:
Use of effective contraception | 4 months
  The proportion reporting current use of effective contraception (pill, intrauterine device, injection, implant, patch)
Acceptability of individual effective contraceptive methods | 4 months
  The proportion reporting that individual methods of effective contraception are acceptable (pill, intrauterine device, injection, implant, patch)
Discontinuation of effective contraception | 4 months
  The proportion reporting use of effective contraception at any time during the 4 months (pill, intrauterine device, injection, implant, patch)
Service uptake | 4 months
  The proportion reporting attending a sexual health service during the 4 months
Unintended pregnancy | 4 months
  The proportion reporting that they became pregnant and did not want to become pregnant during the study
Induced abortion | 4 months
  The proportion reporting having an abortion during the study

OTHER OUTCOMES:
Knowledge of effective contraception | 4 months
  Score on the knowledge measure
Perceived norms in relation to using and communicating with partners about contraception | 4 months
  Responses to the perceived norms scales
Personal agency in using and communicating with partners about contraception | 4 months
  Responses to the personal agency scales
Intention to use effective contraception | 4 months
  Response to the intention scale
Intervention 'dose' received | 4 months
  If participants read all, some, most or none of the messages and if they stopped the messages

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Free, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Palestinian Family Planning and Protection Association, Jerusalem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] McCarthy OL, Zghayyer H, Stavridis A, Adada S, Ahamed I, Leurent B, Edwards P, Palmer M, Free C. A randomized controlled trial of an intervention delivered by mobile phone text message to increase the acceptability of effective contraception among young women in Palestine. Trials. 2019 Apr 23;20(1):228. doi: 10.1186/s13063-019-3297-4. PMID 31014358
- [Derived] McCarthy OL, Wazwaz O, Jado I, Leurent B, Edwards P, Adada S, Stavridis A, Free C. An intervention delivered by text message to increase the acceptability of effective contraception among young women in Palestine: study protocol for a randomised controlled trial. Trials. 2017 Oct 3;18(1):454. doi: 10.1186/s13063-017-2191-1. PMID 28974258